CLINICAL TRIAL: NCT05499481
Title: Short Against Long Antibiotic Therapy for Infected Orthopedic Sites
Acronym: SALATIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2022-01012
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Devices Associated With Misadventures; Infection, Surgical Site; Antibiotic Side Effect
Keywords: Orthopedic infectionsT; Duration; Antibiotic Therapy; Randomized-Controlled Trial
MeSH Terms: conditions — Surgical Wound Infection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: The investigators will perform two concomitant RCTs, depending on the presence of infected osteosynthesis material at enrolment:
  - SALATIO 1. Infected implant not removed (or new material inserted): Randomization 6 vs. 12 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.
  - SALATIO 2. Infected implant without residual material (definitive removal or within the interval of a two-stage exchange): Randomization 3 vs. 6 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Antibiotic Arm (Active Comparator): Without implant material in place:
  6 weeks of systemic post-surgical antibiotic therapy
  With mateial in place 12 weeks of systemic post-surgical antibiotic therapy
  Interventions: Drug: Antibiotic
- Short Antibiotic Arm (Experimental): Without implant material in place:
  3 weeks of systemic post-surgical antibiotic therapy
  With mateial in place 6 weeks of systemic post-surgical antibiotic therapy
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — The investigators will perform two concomitant RCTs, depending on the presence of infected osteosynthesis material at enrolment:
  - SALATIO 1. Infected implant not removed (or new material inserted): Randomization 6 vs. 12 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.
  - SALATIO 2. Infected implant without residual material (definitive removal or within the interval of a two-stage exchange): Randomization 3 vs. 6 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.

SUMMARY:
The investigators will perform two concomitant RCTs, depending on the presence of infected osteosynthesis material at enrolment:

- SALATIO 1. Infected implant not removed (or new material inserted): Randomization 6 vs. 12 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.

- SALATIO 2. Infected implant without residual material (definitive removal or within the interval of a two-stage exchange): Randomization 3 vs. 6 weeks (+/- 5 days) of total antibiotic therapy counted since the first debridement for infection. Early switch to oral targeted therapy.

DETAILED DESCRIPTION:
The optimal duration of postoperative, systemic antibiotic therapy for implant-related orthopedic infections, with or without implant removal, is unknown.

Retrospective studies suggest that a maximum duration of 6 weeks is not inferior to longer administrations; even if the infected implants are kept in place or during a one-stage exchange. Prospective-randomized trials (RCT) suggest that even shorter durations, such 3 or 4 weeks, are possible, when the implant is removed. Likewise, in prospective studies, 6 or 8 weeks of systemic antibiotics are not inferior to the current 12 weeks during DAIR (debridement, antibiotic and implant retention), or during the one-stage exchange; except for one single RCT suggesting a better outcome for 12 weeks in the substrata of arthroplasty infections undergoing the DAIR procedure.

However, these RCTs concern selected branches of orthopedic surgery; especially prosthetic joint infections. The investigators intend to expand these evaluations to all fields of orthopedic and hand surgery. The only exceptions would be spine surgery, for which a multicenter, separate RCT is already under way (SASI-trials). The second exception would be the treatment of implant-free diabetic foot infections, for which two RCTs are underway.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years on admission
* Orthopedic bone and implant infections including musculoskeletal grafts
* Intraoperative debridement with any surgical technique
* 12 months of scheduled follow-up from hospitalization
* Bacterial orthopedic infections of any nature
* First or second episode of infection

Exclusion Criteria:

* Mycobacterial, fungal, nocardial, and Actinomyces infections
* Purely soft tissue infections
* Non-resected cancer in the infection site
* Purely intrasynovial infections (native joint septic arthritis)
* More than three debridements performed for infection
* Absence of at least one surgical intraoperative debridement
* Spine infections (investigated in another trial)10
* Diabetic foot infections (investigated in another trial)7
* Documented endocarditis according to the Duke criteria
* At least 2 prior infection episodes at the actual infection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical remission related to the duration of total, postdebridement, antibiotic use | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  Clinical assessment during routine surgical controls. Definition of clinical failure accoding to to sandard criteria in the literature (surgical revision, pain, local inflammation, discharge, several deep intraoperative bacterial tissue samples)
Microbiological recurrence in relation to the total, postdebridement, antibiotic use | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  Recurrence of infection, with the same pathogens, after completing the antibiotic treatment for the index infection

SECONDARY OUTCOMES:
Description of all clinical failures of any sort | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  Need for hospitalisation or revision surgery for any non-infectious failures related to the operation wound (hematoma, seroma, internal (closed) fractures, dislocation of implants)
Adverse events in each study arm, and in relation to the antibiotics used | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  All adverse events during the therapy and follow-up time , with an emphasis on antibiotic-related adverse events (according to medical judgement). Numbers and descriptions.
Length of hospital stay in acute care surgery (without rehabilitation) | 6 weeks postoperatively, or 1 year postoperatively in case of implant-related orthopedic surgery
  The duration of the hospital stay for every episode in both randomizing arm

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, Professor, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators might share anonymized key elements upon reasonable scientific request to the corresponding persons
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after the first interim analysis
Access Criteria: The investigators might share anonymized key elements upon reasonable scientific request to the corresponding persons

REFERENCES:
- [Background] Chaussade H, Uckay I, Vuagnat A, Druon J, Gras G, Rosset P, Lipsky BA, Bernard L. Antibiotic therapy duration for prosthetic joint infections treated by Debridement and Implant Retention (DAIR): Similar long-term remission for 6 weeks as compared to 12 weeks. Int J Infect Dis. 2017 Oct;63:37-42. doi: 10.1016/j.ijid.2017.08.002. Epub 2017 Aug 10. PMID 28804007
- [Background] Bernard L, Legout L, Zurcher-Pfund L, Stern R, Rohner P, Peter R, Assal M, Lew D, Hoffmeyer P, Uckay I. Six weeks of antibiotic treatment is sufficient following surgery for septic arthroplasty. J Infect. 2010 Jul;61(2):125-32. doi: 10.1016/j.jinf.2010.05.005. Epub 2010 Jun 9. PMID 20540962
- [Background] Hirsiger S, Betz M, Stafylakis D, Gotschi T, Lew D, Uckay I. The Benefice of Mobile Parts' Exchange in the Management of Infected Total Joint Arthroplasties with Prosthesis Retention (DAIR Procedure). J Clin Med. 2019 Feb 9;8(2):226. doi: 10.3390/jcm8020226. PMID 30744128
- [Background] Farhad R, Roger PM, Albert C, Pelligri C, Touati C, Dellamonica P, Trojani C, Boileau P. Six weeks antibiotic therapy for all bone infections: results of a cohort study. Eur J Clin Microbiol Infect Dis. 2010 Feb;29(2):217-22. doi: 10.1007/s10096-009-0842-1. Epub 2009 Dec 10. PMID 20012334
- [Background] Gariani K, Pham TT, Kressmann B, Jornayvaz FR, Gastaldi G, Stafylakis D, Philippe J, Lipsky BA, Uckay L. Three Weeks Versus Six Weeks of Antibiotic Therapy for Diabetic Foot Osteomyelitis: A Prospective, Randomized, Noninferiority Pilot Trial. Clin Infect Dis. 2021 Oct 5;73(7):e1539-e1545. doi: 10.1093/cid/ciaa1758. PMID 33242083
- [Background] Waibel F, Berli M, Catanzaro S, Sairanen K, Schoni M, Boni T, Burkhard J, Holy D, Huber T, Bertram M, Laubli K, Frustaci D, Rosskopf A, Botter S, Uckay I. Optimization of the antibiotic management of diabetic foot infections: protocol for two randomized controlled trials. Trials. 2020 Jan 8;21(1):54. doi: 10.1186/s13063-019-4006-z. PMID 31915048
- [Background] Benkabouche M, Racloz G, Spechbach H, Lipsky BA, Gaspoz JM, Uckay I. Four versus six weeks of antibiotic therapy for osteoarticular infections after implant removal: a randomized trial. J Antimicrob Chemother. 2019 Aug 1;74(8):2394-2399. doi: 10.1093/jac/dkz202. PMID 31106353
- [Background] Rod-Fleury T, Dunkel N, Assal M, Rohner P, Tahintzi P, Bernard L, Hoffmeyer P, Lew D, Uckay I. Duration of post-surgical antibiotic therapy for adult chronic osteomyelitis: a single-centre experience. Int Orthop. 2011 Nov;35(11):1725-31. doi: 10.1007/s00264-011-1221-y. Epub 2011 Feb 12. PMID 21318568
- [Background] Betz M, Uckay I, Schupbach R, Grober T, Botter SM, Burkhard J, Holy D, Achermann Y, Farshad M. Short postsurgical antibiotic therapy for spinal infections: protocol of prospective, randomized, unblinded, noninferiority trials (SASI trials). Trials. 2020 Feb 6;21(1):144. doi: 10.1186/s13063-020-4047-3. PMID 32028985
- [Background] Argenson JN, Arndt M, Babis G, Battenberg A, Budhiparama N, Catani F, Chen F, de Beaubien B, Ebied A, Esposito S, Ferry C, Flores H, Giorgini A, Hansen E, Hernugrahanto KD, Hyonmin C, Kim TK, Koh IJ, Komnos G, Lausmann C, Loloi J, Lora-Tamayo J, Lumban-Gaol I, Mahyudin F, Mancheno-Losa M, Marculescu C, Marei S, Martin KE, Meshram P, Paprosky WG, Poultsides L, Saxena A, Schwechter E, Shah J, Shohat N, Sierra RJ, Soriano A, Stefansdottir A, Suleiman LI, Taylor A, Triantafyllopoulos GK, Utomo DN, Warren D, Whiteside L, Wouthuyzen-Bakker M, Yombi J, Zmistowski B. Hip and Knee Section, Treatment, Debridement and Retention of Implant: Proceedings of International Consensus on Orthopedic Infections. J Arthroplasty. 2019 Feb;34(2S):S399-S419. doi: 10.1016/j.arth.2018.09.025. Epub 2018 Oct 19. No abstract available. PMID 30348550
- [Background] Lora-Tamayo J, Euba G, Cobo J, Horcajada JP, Soriano A, Sandoval E, Pigrau C, Benito N, Falgueras L, Palomino J, Del Toro MD, Jover-Saenz A, Iribarren JA, Sanchez-Somolinos M, Ramos A, Fernandez-Sampedro M, Riera M, Baraia-Etxaburu JM, Ariza J; Prosthetic Joint Infection Group of the Spanish Network for Research in Infectious Diseases-REIPI. Short- versus long-duration levofloxacin plus rifampicin for acute staphylococcal prosthetic joint infection managed with implant retention: a randomised clinical trial. Int J Antimicrob Agents. 2016 Sep;48(3):310-6. doi: 10.1016/j.ijantimicag.2016.05.021. Epub 2016 Aug 3. PMID 27524103
- [Background] Bernard L, Arvieux C, Brunschweiler B, Touchais S, Ansart S, Bru JP, Oziol E, Boeri C, Gras G, Druon J, Rosset P, Senneville E, Bentayeb H, Bouhour D, Le Moal G, Michon J, Aumaitre H, Forestier E, Laffosse JM, Begue T, Chirouze C, Dauchy FA, Devaud E, Martha B, Burgot D, Boutoille D, Stindel E, Dinh A, Bemer P, Giraudeau B, Issartel B, Caille A. Antibiotic Therapy for 6 or 12 Weeks for Prosthetic Joint Infection. N Engl J Med. 2021 May 27;384(21):1991-2001. doi: 10.1056/NEJMoa2020198. PMID 34042388
- [Derived] Zendeli F, Jedrusik A, Schaefer RO, Albrecht D, Betz M, Waibel FWA, Grober T, Kuhne N, Konneker S, Uckay I. Pathogen-Specific Risk for Iterative Surgical Debridement in Orthopedic Infections: A Prospective Multicohort Analysis. J Clin Med. 2025 Dec 10;14(24):8750. doi: 10.3390/jcm14248750. PMID 41464652
- [Derived] Uckay I, Wirth S, Zorner B, Fucentese S, Wieser K, Schweizer A, Muller D, Zingg P, Farshad M. Study protocol: short against long antibiotic therapy for infected orthopedic sites - the randomized-controlled SALATIO trials. Trials. 2023 Feb 18;24(1):117. doi: 10.1186/s13063-023-07141-2. PMID 36803837